CLINICAL TRIAL: NCT05582772
Title: TOward a comPrehensive Supportive Care Intervention for Older Men With Metastatic Prostate Cancer (TOPCOP3): a Pilot RCT and Process Evaluation
Brief Title: TOward a comPrehensive Supportive Care Intervention for Older Men With Metastatic Prostate Cancer
Acronym: TOPCOP3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 4090
Record Dates: First submitted 2022-09-16; First posted 2022-10-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Prostate Cancer
Keywords: Geriatric assessment; ARAT; Supportive Care; Older men
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Geriatric Assessment; Therapeutics

STUDY DESIGN:
Intervention Model Description: This model will provide within-group change scores for both co-primary outcomes (i.e., grade 3-5 toxicity and QOL) along with standard deviations and responsiveness measure. These data will guide selection of the single or dual primary outcome for the definitive phase III RCT as well as inform sample size calculations. Importantly, they will not be used to determine the clinically important difference used to plan for the phase III RCT. These 2 co-primary outcomes were selected based on literature review, clinical input, and patient-partner input.
Masking Description: Given the nature of the intervention, it is not possible to blind patients or the project team to allocation, however, the statistician is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- GA+M Intervention (Active Comparator): GA+M intervention arm All participants in the GA+M intervention arm will undergo a standardized GA by a trained nurse and geriatrician. The GA will include 8 domains (comorbidity, medication review, function, falls risk, nutrition, social supports, cognition, and mood) similar to our 5C protocol.
  Based on any detected abnormalities or issues, a standardized set of strategies will be implemented (e.g. increased falls risk will lead to detailed assessment of balance and gait, consideration of gait aid, and referral to outpatient physiotherapy). This follows the standard approach to implementing GA similar to recent trials in geriatric oncology including 5C. Telephone follow-ups at 1, 3 and 6 months by the nurse and review with the geriatrician as needed will be done to ensure identified issues have been addressed.
  Interventions: Other: GA+M Intervention
- RSM Intervention (Active Comparator): RSM Intervention All participants in the RSM intervention arm will receive once-weekly symptom monitoring via email-based surveys using the 9-item Edmonton Symptom Assessment Scale within a secure customized REDCap interface. If patients prefer, weekly telephone calls will be done instead by a research assistant to elicit If there are moderate or severe symptoms (score of 4+ out of 10), an oncology nurse will obtain more detailed symptom information and provide evidence-based symptom-targeted recommendations using the pan-Canadian Oncology Symptom Triage and Remote Support (COSTaRS) Practice Guide. Symptom monitoring will continue for 6 months or discontinuation of treatment.
  Interventions: Other: RSM intervention
- GA+RSM intervention (Active Comparator): GA+RSM Combination Participants will receive both strategies as detailed above, with a GA at baseline.
  Interventions: Other: GA+RSM intervention
- Control (No Intervention): Control Usual care consists of brief verbal education and a drug pamphlet to all patients when starting an ARAT. There is no GA+M and no RSM at either site. Patients have access to a 24x7 oncology nursing line or a 24/7 pharmacy line.

INTERVENTIONS:
Other: GA+M Intervention — Typically 8 domains (cognition, comorbidities, falls risk, functional status, medication use, mood - depression, nutritional status, social support) are examined by a team consisting of a nurse and geriatrician. A GA has multiple benefits and has been recommended for all older adults considering chemotherapy by the American Society of Clinical Oncology (ASCO). For a GA to be most useful it needs to be followed by co-management of identified issues.
  Other Names: Geriatric assessment and management
  Arms: GA+M Intervention
Other: RSM intervention — Telephone-based, symptom management of patients with cancer
  Other Names: Remote symptom monitoring
  Arms: RSM Intervention
Other: GA+RSM intervention — Combining a geriatric assessment and remote symptom control
  Other Names: Geriatric assessment and remote symptom monitoring
  Arms: GA+RSM intervention

SUMMARY:
TOPCOP3 is a pilot factorial RCT of geriatric assessment and management, remote symptom monitoring, both interventions or neither, accompanied by an embedded process evaluation. This design is widely used to guide the evaluation of complex interventions and provides important data to aid design of larger RCTs. The trial itself falls within pilot trial goals including obtaining variance estimates for outcomes, assessment of recruitment potential, and understanding implementation issues vital to designing a larger trial. The investigators have clear feasibility objectives and an analytic plan as well as criteria to determine success and strong support from cancer advocacy and policy groups.

DETAILED DESCRIPTION:
Emerging data from supportive care intervention trials in people receiving chemotherapy suggest 2 different approaches - geriatric assessment and management (GA+M) and remote symptom monitoring (RSM) - may be associated with improved time on treatment, improved QOL, reduced toxicity, reduced unplanned health care use, and possibly prolonged overall survival. These 2 interventions have not been tested in combination or in people receiving treatments other than chemotherapy (such as ARATs). This RCT includes an embedded process evaluation of GA+M and RSM versus usual care to gather key efficacy and implementation data needed to design a definitive phase III RCT.

The next logical step in our research program is an intervention examining GA+M, RSM, or the combined intervention to improve the health and treatment tolerability for older men with mPC on ARATs. The pilot trial will gather key clinical outcome and feasibility data needed to inform a definitive phase III RCT; a necessary step in providing clinicians a greatly needed evidence-based supportive care intervention. The intervention was designed in partnership with patients and knowledge users, which will result in more relevant findings and greater health impact.

A total of 168 patients will be enrolled in the RCT across 2 centres. Based on TOPCOP1 and TOPCOP2, both of which included the two centres in TOPCOP3, the recruitment rate was 2-3 patients per week. There are 3-5 eligible patients per week across the two sites. Assuming a conservative recruitment rate of 50%, the investigators expect recruitment for this study to take 18 months.

Randomization will be centralized using REDCap, a secure web-based electronic data entry system. Patients will be allocated in a 1:1:1:1 ratio to GA+M, RSM, combined, or control, with stratification by mPC subtype (castration-sensitive or resistant) following recommended guidelines on number of strata. Permuted blocks of variable size will be used.

Given the nature of the intervention, it is not possible to blind patients or the project team to allocation. However, participants will be randomized, allocation will be concealed, variable permuted blocks will be used, 1 of the 2 co-primary outcomes will be assessed by blinded assessors (toxicity), validated measures will be used, several outcomes will be verified by independent data collection (treatment toxicity, overall survival), and the trial statistician will be blinded during the trial and during analysis of the main study results, similar to our 5C trial.

GA+M intervention arm:

All participants in the GA+M intervention arm will undergo a standardized GA by a trained nurse and geriatrician. The GA will include 8 domains (comorbidity, medication review, function, falls risk, nutrition, social supports, cognition, and mood) similar to our 5C protocol.

Based on any detected abnormalities or issues, a standardized set of strategies will be implemented (e.g. increased falls risk will lead to detailed assessment of balance and gait, consideration of gait aid, and referral to outpatient physiotherapy). This follows the standard approach to implementing GA similar to recent trials in geriatric oncology including 5C.Telephone follow-ups at 1, 3 and 6 months by the nurse and review with the geriatrician as needed will be done to ensure identified issues have been addressed.

RSM Intervention arm:

All participants in the RSM intervention arm will receive once-weekly symptom monitoring via email-based surveys using the 9-item Edmonton Symptom Assessment Scale within a secure customized REDCap interface. If patients prefer, weekly telephone calls will be done instead by a research assistant to elicit symptoms. In our prior study, almost half the participants preferred telephone calls. If there are moderate or severe symptoms (score of 4+ out of 10), an oncology nurse will obtain more detailed symptom information and provide evidence-based symptom-targeted recommendations using the pan-Canadian Oncology Symptom Triage and Remote Support (COSTaRS) Practice Guide. For moderate symptoms that persist even after follow up, if the RSM nurse feels that the patient is clinically stable in the same symptom based on at least 2 phone assessments, 1 week apart, and there are no further COSTaRS-directed interventions to be implemented for this symptom based on the RSM nurse's judgement the following silencing protocol can be adopted: The RSM nurse will inform the study coordinator to not flag the study nurse for further moderate alerts for the same symptom if the score is identical to the prior week (i.e. to silence the alarm). If the score changes from moderate to severe, or increases 2 points within the same verbal descriptor severity category (e.g. 4 to 6/10, both are moderate) then the nurse is alerted again. The silencing option will remain for 4 weeks then expire. Symptom monitoring will continue for 6 months or discontinuation of treatment (whichever comes first). If treatment is discontinued for a period of 3 weeks, the weekly ESAS questionnaire will not be sent out to the participant until treatment is resumed. An escalation protocol will also be followed for persistent symptoms or those deemed out of scope for nurse-guided self-management, with referral to the patient's oncologist or urgent care as appropriate. Oncology nurses are ideally situated to be the primary point of contact with oncology patients, can promote patient self-efficacy, provide counselling and support, and can handle 87% of issues without needing physician input.

GA+RSM Combination:

Participants will receive both strategies as detailed above, with a GA at baseline.

Control:

Usual care consists of brief verbal education and a drug pamphlet to all patients when starting an ARAT. There is no GA+M and no RSM at either site. Patients have access to a 24x7 oncology nursing line.

Patients will receive the TOPCOP3 intervention for a duration of 6 months. This balances participant burden and resources with a timeframe that is sufficient to observe clinical and implementation outcomes (most severe toxicity is observed within the first 3 months of treatment. Most GA+M trials have been 6 months in duration.

ELIGIBILITY:
Inclusion Criteria:

1. Starting an ARAT or started an ARAT within 2 weeks prior to being approached or switching ARATs due to progression or toxicity
2. Diagnosed with mPC (castration-sensitive or resistant) or nmCRPC (non-metastatic castration-resistant prostate cancer)
3. At least 65 years old
4. Able to provide written informed consent
5. Has a working telephone

Exclusion Criteria:

1. Unable to speak English (as contact with the nurse interventionist is via phone, not all outcome measures are available in multiple languages)
2. Major neuropsychiatric abnormalities (severe depression or moderate-severe dementia)
3. Life expectancy <3 months as estimated by the oncologist

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — This RCT is in metastatic prostate cancer, which occurs in men only.
Enrollment: 168 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Grade 3-5 Toxicity | 6 months
  Grade 3-5 toxicity. This will be coded as at least one grade 3-5 toxicity vs none, measured based on review of clinical notes supplemented by interviews with patients by trained research staff and verified by a blinded physician. Toxicities will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Health related quality of life in patients with metastatic prostate cancer | 6 months
  QOL will be measured by patient self-report using the EQ-5D-5L, which is the EuroQol 5 dimensions of health questionnaire. This is a widely used, psychometrically valid brief generic QOL questionnaire.

SECONDARY OUTCOMES:
Number of patients with treatment discontinuation | 6 months
  Early treatment discontinuation due to toxicity. This will be based on chart review and oncologist clarification.
Number of patients with treatment modification | 6 months
  Treatment modification after GA (change in ARAT dose/agent). Based on chart review. For GA+M arms only
Number of patients with severe symptoms | 6 months
  Symptom severity. This is measured using the 15-item Symptom Distress Scale. This is a patient reported outcome (PRO).
Number of patients with decline in Instrumental Activities of Daily Living (IADL) | 6 months
  Decline in IADL using the Older Adults Resources and Services (OARS) scale. This is a patient reported outcome (PRO).
Number of patients with unplanned health care | 6 months
  Unplanned health care use. Emergency room visits and hospital admissions will be recorded at each time point with a combination of patient interviews and electronic health record audit
Fatigue | 6 months
  Fatigue - measured using the Brief Fatigue Inventory (BFI). This is a patient reported outcome (PRO).
Insomnia | 6 months
  Insomnia will be measured using the Insomnia Severity Index. This is a patient reported outcome (PRO).
Anorexia and cachexia | 6 months
  Anorexia and Cachexia is measured with the Functional Assessment of Anorexia-Cachexia Therapy scale (Functional Assessment of Anorexia/Cachexia FAACT-A/CS-12). This is a patient reported outcome (PRO).
Depression | 6 months
  Depression will be measured using the 9-item Patient Health Questionnaire (PHQ-9). This is a patient reported outcome (PRO).

OTHER OUTCOMES:
Process evaluation: Feasibility | 6 months
  The trial will be determined to be feasible if recruitment rate is 60% or higher, retention rate is 85% or higher, adherence is 90% or higher, outcome capture is 90% or higher, and contamination rate is 5% or less.
Process evaluation: Acceptability | 6 months
  Likert scale satisfaction survey.

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Alibhai, MD, Principal Investigator — UHN - Princess Margaret Cancer Centre
Locations (3):
- Canada (3):
  - St. Michael's hospital, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alibhai SMH, Puts M, Jin R, Godhwani K, Antonio M, Abdallah S, Feng G, Krzyzanowska MK, Soto-Perez-de-Celis E, Papadopoulos E, Mach C, Nasiri F, Sridhar SS, Glicksman R, Moody L, Bender J, Clarke H, Matthew A, McIntosh D, Klass W, Emmenegger U. TOward a comPrehensive supportive Care intervention for Older men with metastatic Prostate cancer (TOPCOP3): A pilot randomized controlled trial and process evaluation. J Geriatr Oncol. 2024 Jul;15(6):101750. doi: 10.1016/j.jgo.2024.101750. Epub 2024 Mar 23. PMID 38521641